CLINICAL TRIAL: NCT03550924
Title: Increasing Duration of Apnea Without Desaturation at Induction of Anesthesia in Morbidly Obese Patients Using "Transnasal Humidified Rapid Insufflation Ventilatory Exchange (THRIVE)"
Brief Title: Transnasal Humidified Rapid Insufflation Ventilatory Exchange in Morbidly Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Hamp, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2270/2017
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia Intubation Complication; Anesthesia

STUDY DESIGN:
Intervention Model Description: Prospective, single center, randomized, observer blinded, controlled
Who Masked: Investigator
Masking Description: The monitor measuring the main outcome parameter will be in a separate room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low flow Oxygen Group (Active Comparator): low flow passive oxygenation during laryngoscopy with 10l/min oxygen via standard nasal prongs
  Interventions: Procedure: low flow passive oxygenation
- THRIVE Group (Experimental): high flow passive oxygenation during laryngoscopy with 120l/min oxygen via THRIVE system
  Interventions: Procedure: high flow passive oxygenation

INTERVENTIONS:
Procedure: low flow passive oxygenation — low flow passive oxygenation during laryngoscopy with 10l/min oxygen via standard nasal prongs
  Arms: Low flow Oxygen Group
Procedure: high flow passive oxygenation — high flow passive oxygenation during laryngoscopy with 120l/min oxygen via THRIVE system
  Arms: THRIVE Group

SUMMARY:
This project will investigate the duration of apnea without desaturation when using transnasal humidified rapid insufflation ventilatory exchange (THRIVE) vs. low flow nasal oxygen at anesthesia induction in obese patients.

DETAILED DESCRIPTION:
Background Providing safe anesthesia for surgery in obese patients requires specific consideration of the pathophysiological changes and respiratory complications are frequent. Anesthesia induction needs special attention in this patient population. A decrease in functional residual capacity (FRC) after induction of anesthesia dramatically shortens the duration of apnea without desaturation (DAWD) during which the airway can be secured.

Several measures such as positioning in a semi sitting position, preoxygenation with PEEP and passive insufflation of oxygen during laryngoscopy have been shown to prolong the DAWD. None of these measures is able to produce positive endexpiratory pressure (PEEP) during laryngoscopy which would counteract the loss of FRC and therefore prolong the DAWD further.

Transnasal humidified rapid insufflation ventilator exchange (THRIVE, also knowns as "high flow nasal oxygen therapy" and "heated and humidified nasal oxygen") devices have been used for several years in intensive care and are available from numerous vendors. With THRIVE, heated and humidified oxygen is insufflated via nasal prongs at a rate up to 120 l/minute and it has been shown that this creates levels of PEEP, proportional to the amount of gas flow. Using THRIVE during the apneic phase of anesthesia induction in obese patients might be superior compared to low flow oxygen techniques as THRIVE generates PEEP during laryngoscopy, which might counteract the loss of FRC and consequently might prolong the DAWD.

Aim of the project This project will investigate the DAWD when using THRIVE vs. low flow nasal oxygen at anesthesia induction in obese patients.

Hypothesis The duration of apnea without desaturation is longer in the "THRIVE" group compared to the "low flow oxygen" group.

Methods The study will be conducted as a single center, prospective, randomized, controlled trial at the Medical University of Vienna, Austria.

Forty adult patients of the ASA classification 2 and 3 with a BMI >40 undergoing elective surgery under general anesthesia will be included. Patients with expected difficult airway, patients with an oxygen saturation <98% despite preoxygenation, patients with nasal obstruction, smokers (>10 cigarettes/day), patients with chronic respiratory disease, patients unable to give consent, and pregnant or breastfeeding patients will be excluded.

Patients will be randomly assigned to one of two groups ("low flow oxygen" or "THRIVE" group) and anesthesia will be induced in a standardized fashion in both groups. During laryngoscopy, patients in the low flow group will receive nasal oxygen insufflation at a rate of 10 l/min and patients in the THRIVE group will receive oxygen at a rate of 120 l/min via a THRIVE system. Difficult laryngoscopy will be simulated and intubation will be performed as soon as oxygen saturation drops to 95%. The time from anesthesia induction until oxygen saturation drops to 95% (DAWD) will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* American Society of Anesthesiologists physical status classification class 2-3
* BMI > 40
* elective surgery under general anesthesia

Exclusion Criteria:

* expected difficult airway (El Ganzouri Risk Index > 6)
* oxygen saturation of less than 98% despite adequate preoxygenation,
* nasal obstruction
* smoker, more than 10 cigarettes per day
* chronic respiratory disease
* FEV1 (forced expiratory volume in one second) < 70%
* elevated intracranial pressure
* unable to give informed consent
* Pregnant or breast feeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Duration of safe apnea | duration from the application of rocuronium until the oxygen saturation drops to 95% during laryngoscopy or a maximum of 15 minutes if the oxygen saturation does not drop to this level.
  The duration until oxygen saturation drops to 95% during laryngoscopy

SECONDARY OUTCOMES:
blood gas analysis | every 2 minutes after rocuronium was given until 2 minutes after intubation
  arterial blood samples will be taken every 2 minutes after rocuronium was given until 2 minutes after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hamp, Doctor, Principal Investigator — Department of Anaesthesia and Intensive Care Medicine
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided